CLINICAL TRIAL: NCT06167551
Title: The Effect of 3 Different Auditory Applications on Pain, Crying Duration and Physiological Parameters During Newborn Heel Prick Procedures
Brief Title: The Effect of 3 Different Auditory Applications on Newborn Heel Prick Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Zeynem YILDIRIM BALKAN, Dr. Lecturer and Principal Investigator, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TNKU-Z.BALKAN-1
Record Dates: First submitted 2023-10-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Newborn Pain
Keywords: newborn; heel prick; music; pain care

STUDY DESIGN:
Intervention Model Description: Comparison of 3 different auditory applications with the control group during heel prick collection in newborns.
Who Masked: Participant, Outcomes Assessor
Masking Description: The baby's crying time will be monitored and recorded. KTA and SpO2 will be recorded by the researcher during blood collection. Pain assessment of the babies will be made by two independent neonatal nurses other than the researcher. Both observers must have worked in the clinic for at least 5 years.
  Analysis of the data will be done by an independent analyst, not by researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mother lullaby group (Experimental): group listening to mother's lullaby
  Interventions: Other: mother lullaby group
- white noise group (Experimental): group listening to white noise
  Interventions: Other: white noise group
- classical music group (Experimental): group listening to classical music
  Interventions: Other: classical music group
- Control group (Other): No intervation
  Interventions: Other: Contol Group

INTERVENTIONS:
Other: mother lullaby group — mother's lullaby: the mother will be made to sing her own lullaby 5 minutes before the heel prick.
  Arms: mother lullaby group
Other: white noise group — white noise: 5 minutes before taking heel prick blood, white noise will be started to be played on an MP3 player with white noise. The MP3 player will be placed in the crib where the baby lies, at the baby's bedside, at least 20 cm away from the baby's head. After the MP3 player is turned on, the sound level will be measured at the baby's ear level with a decibel meter and adjusted so that it does not exceed 70 decibels.
  Arms: white noise group
Other: classical music group — classical music: 5 minutes before heel prick, classical music will be started to be played from the MP3 player with white noise. The MP3 will be placed inside the crib where the baby lies, at the baby's bedside, at least 20 cm away from the baby's head. After the MP3 player is turned on, the sound level will be measured at the baby's ear level with a decibel meter and adjusted so that it does not exceed 70 decibels.
  Arms: classical music group
Other: Contol Group — No intervation
  Other Names: No intervation
  Arms: Control group

SUMMARY:
In pain management of neonates in interventional applications, health professionals should be able to evaluate pain, reduce or eliminate pain. Pharmacologic and nonpharmacologic methods are used in pain management. Pharmacological, opioid analgesics, sedatives and local anesthetics are used. Nonpharmacologic methods include breastfeeding, giving pacifiers, oral sucrose, music, massage, therapeutic touch and nesting, positioning such as fetal positioning, wrapping, kangaroo care, rocking and cradling.

Music makes positive changes in oxygen saturation level and peak heart rate values and reduces stress and pain. Classical music with light rhythmic emphasis and steady rhythm accompanied by a simple human voice or a single instrument, music performed by female vocalists (mother's voice, lullabies with female voice) and white noise similar to intrauterine sounds are among the types of music that have a positive effect on newborns.

This study was planned as a randomized controlled experimental design to compare the lullaby, classical music and white noise song by the mother to the newborn before and during heel prick blood collection with the control group and to determine which application gives superior results to the newborn's pain level, crying time and physiological parameters.

DETAILED DESCRIPTION:
In pain management of newborns in interventional applications, health professionals should be able to evaluate pain and reduce or eliminate pain. Pharmacological and non-pharmacological methods are used in the management of pain. Non-pharmacological methods: practices such as breastfeeding, giving a pacifier, giving oral sucrose, listening to music, massage, therapeutic touching and nesting, positioning the fetus such as wrapping, giving kangaroo care, rocking and holding.

The newborn's response to sound often leads to changes in breathing and heart rate. Mild to moderate sounds (55-75 dB), such as speech and music, cause a decrease in heart rate and create an orientation response. Music makes positive changes in oxygen saturation level and heart rate peak values, and also reduces stress and pain. Arnon et al. determined that letting newborns in intensive care listen to music has a positive effect on reducing pain and anxiety, making it easier for newborns to fall asleep and increasing their sleep quality. Classical music with a light rhythmic emphasis and constant rhythm accompanied by a simple human voice or a single instrument, music performed by female vocalists (mother's voice, lullabies with a female voice) and white noise similar to intrauterine sounds are among the types of music that have a positive effect on newborns.

Heel prick pricking in newborns causes pain, which results in increased blood pressure and pulse rate, decreased SpO2, and crying. For this reason, this study was designed as a randomized controlled experimental design to compare the classical music and white noise and lullaby applications to the newborn before and during heel blood collection with the control group and to determine which application provides superior results on the newborn's pain level, crying duration and physiological parameters.

Research Purpose and Type This research was planned as a randomized controlled experimental design to compare the lullaby, classical music and white noise aplications to the newborn during the heel prick prick procedure with the control group.

Research Variables Independent variables; Lullaby your mother sings, white noise, classical music Dependent variables; Heart rate peak (HRV), oxygen saturation (SpO2), NIPS score, NIAPAS score, crying duration.

Place and Time to Conduct the Research The research will be carried out between February 2024 and June 2024 in the Neonatal Intensive Care Unit of Gaziantep Cengiz Gökçek Gynecology and Children's Hospital.

The population of the research It will create term newborns born at 38-42 weeks of gestation in the Neonatal Intensive Care Unit of Gaziantep Cengiz Gökçek Gynecology and Children's Hospital between February 2024 and June 2024. Postpartum 24-72. These are the newborns whose heel blood will be taken during Sample; The sample number of the study was determined by power analysis. The thesis study, which evaluated the effect of different auditory interventions on pain in heel blood collection in newborns, was taken as an example. According to the NIPS pain assessment scale used in the study, the average score of the results during the procedure was 4.26±2.16 in the 1st experimental group, 4.81±2.18 in the 2nd experimental group, 5.02±2.00 in the 3rd experimental group, and 5.93±1.32 in the control group. In this study, it was anticipated that the NIPS score average difference would have a large effect size (.95 large effect), with a 5% alpha margin of error (two-sided) and 80% power, and in the calculation of the number of samples made in the G*Power (3.1.9.2.) program, each It was determined that 20 babies should be included in a group, 80 babies in total. Considering that there may be sample loss for any reason during the research, the aim is to reach 96 newborns (24 babies in each group) by increasing the number of babies by 20% and using statistical parametric analysis methods.

The sample will be randomly selected from the study population. In the study, randomization will be performed using the URN method, which is considered equivalent to the full randomization method. Although this method is shown as UD, it includes two parameters, α and β. These represent balls of two different colors (for example: red and white). α can be white or red, while β will be the exact opposite of the chosen ball colour. One of the balls is chosen randomly, and if the selected ball is white, the subject is assigned to the α group, and if it is red, the subject is assigned to the β group. This selection process is repeated to determine which group the subject will be in.

In the research, the red ball will be the mother's lullaby (intervention group 1), the yellow ball will be white noise (intervention group 2), the blue ball will be classical music (intervention group 3), and the white ball will be the control group. When there is a baby in the clinic that meets the sample selection conditions, these balls prepared by the researcher will be placed in an invisible, dark-colored bag and a random nurse working in the ward will be able to make the selection without seeing it. Which group the baby will be placed in will be determined by the color of the ball coming out of the bag, and the babies will be distributed randomly to the groups.

ELIGIBILITY:
Inclusion Criteria:

* The newborn must be between 38-42 weeks and weigh appropriately for his/her week (Appropriate Gestational Age - AGA),
* Not taking any analgesic, sedative or anticonvulsant medication for at least 6 hours before,
* Feeding at least 1 hour before,
* No fever,
* Not receiving oxygen therapy,
* Not receiving antibiotic treatment
* No congenital anomalies
* Not next to the bed or under the heater
* Not receiving phototherapy,
* Not being connected to a mechanical ventilator

Exclusion Criteria:

* Presence of congenital anomaly,
* Having a chest tube inserted,
* Intracranial bleeding,
* Presence of anomaly that may cause deafness
* Those with a history of epileptic seizures will be excluded.
* The patient's family refuses to participate in the study.

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac apex beat (HRV) | 5 minutes before heel blood collection and at 1, 3 and 5 minutes during heel blood collection.
  HRV will be evaluated before and during heel blood collection. It will be recorded by the researcher during the blood collection process.
Oxygen saturation (SpO2) | 5 minutes before heel blood collection and at 1, 3 and 5 minutes during heel blood collection.
  SpO2 will be evaluated before and during heel blood collection. It will be recorded by the researcher during the blood collection process.
NIPS scale score | NIPS will be evaluated 5 minutes before the heel prick and at 1, 3 and 5 minutes during the heel prick.
  The scale is used to evaluate pain due to procedures performed in term and premature babies. NIPS consists of sections that evaluate 6 behaviors against pain (crying, breathing pattern, arm and leg movements and alertness). Although the total score varies between 0-7, a higher score indicates greater pain intensity.
NIAPAS scale score | NIAPAS will be evaluated 5 minutes before the heel prick and at 1, 3 and 5 minutes during the heel prick.
  NIAPAS scale measures acute pain; It is a scale that includes five behavioral and three physiological indicators given the week of gestation as a contextual factor. As a result of the scoring of the indicators, the score that can be obtained from the scale is between 0-18. Pain intensity is classified as mild pain (0-5), moderate pain (6-9) and severe pain (10-18).
Crying time | The baby's crying time will be 5 minutes before the heel prick and 5 minutes during the heel prick.
  The baby's crying time will be monitored and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Serap BALCI, PHD, Study Director — ISTANBUL UNİVERSİTY CERRAHPAŞA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnon S, Shapsa A, Forman L, Regev R, Bauer S, Litmanovitz I, Dolfin T. Live music is beneficial to preterm infants in the neonatal intensive care unit environment. Birth. 2006 Jun;33(2):131-6. doi: 10.1111/j.0730-7659.2006.00090.x. PMID 16732778
- [Background] Balcı, S. (2006). Beyaz Gürültünün Kolikli Bebeklerde Etkisi. Marmara Üniversitesi Sağlık Bilimleri Enstitüsü Çocuk Sağlığı ve Hastalıkları Hemşireliği Anabilim Dalı. Yüksek Lisans Tezi. İstanbul, Türkiye.
- [Background] Balcı, S., Dur, Ş., Özdemir, Ş., & Kavuncuoğlu, S. (2021). The effect of two different lancets and heel warming on duration of crying and procedure time during blood sampling: A randomized controlled study. Journal of Neonatal Nursing, 27(6), 426-431.
- [Background] Derebent, E., & Yiğit, R. (2008). Yenidoğanda Non-Farmakolojik Ağrı Yönetimi. Fırat Üniversitesi Sağlık Bilimleri Tıp Dergisi, 22(2), 113.
- [Background] Gilad, E., & Arnon, S. (2010). The role of live music and singing as a stress-reducing modality in the neonatal intensive care unit environment. Music and Medicine, 2(1), 18-22
- [Background] Gooding, L. F. (2010). Using music therapy protocols in the treatment of premature infants: An introduction to current practices. The arts in Psychotherapy, 37(3), 211-214
- [Background] İmseytoğlu, D., & Yıldız, S. (2012). YENİDOĞAN YOĞUN BAKIM ÜNİTELERİNDE MÜZİK TERAPİ. Florence Nightingale Journal of Nursing, 20(2), 160-165.
- [Background] Kanbur BN, Mutlu B, Salihoglu O. Validity and reliability of the Neonatal Infant Acute Pain Assessment Scale (NIAPAS) in Turkish: prospective study. Sao Paulo Med J. 2021 Jul-Aug;139(4):305-311. doi: 10.1590/1516-3180.2020.0721.R1.23122020. PMID 34346962
- [Background] Uyar M, Akin Korhan E. [The effect of music therapy on pain and anxiety in intensive care patients]. Agri. 2011 Oct;23(4):139-46. doi: 10.5505/agri.2011.94695. Turkish. PMID 22290677
- [Background] Standley, J. M. (2012). A discussion of evidence-based music therapy to facilitate feeding skills of premature infants: The power of contingent music. The arts in Psychotherapy, 39(5), 379-382.